CLINICAL TRIAL: NCT06467071
Title: Self Help Plus and Post-Migration Living Difficulties Support Intervention: A Randomized Controlled Trial With Syrian Women Under Temporary Protection in Turkey
Brief Title: Self Help Plus and Post-Migration Living Difficulties Support Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Zeynep Keklik, Psychologist, MSc Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH+ZKX2; 0725E271X2 (Other: Istanbul Medipol University)
Record Dates: First submitted 2024-06-09; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Psychological Distress; Psychological Trauma; Mental Health; Refugee Health
Keywords: Syrian Women Refugees; Self Help Plus; Post Migration Living Difficulties
MeSH Terms: conditions — Psychological Trauma; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Help Plus (SH+) combined with a session for Post Migration Living Difficulties (PMLD) (Experimental): The intervention integrates Self Help Plus (SH+) and a session for Post-Migration Living Difficulties (PMLD) for Syrian women. Participants will be randomly assigned to the SH+ combined with the PMLD session (n = 105). The participants in the experimental arm will receive SH+ combined with the PMLD session, by non-specialist facilitators.
  Interventions: Behavioral: SH+ combined with a session for PMLD
- Treatment-As-Usual (TAU) (No Intervention): 105 participants will be randomly allocated to the Treatment as Usual (TAU) group. Mental health services for asylum seekers in Turkey are provided by the Ministry of Health and different non-governmental organizations. These services include psychosocial support, counseling, mental health screenings, and psychotherapy (AIDA, 2020). As usual, treatment includes usual mental health support and assessment following the standard procedures of the Refugees Association Mental Health Unit.

INTERVENTIONS:
Behavioral: SH+ combined with a session for PMLD — The intervention integrates WHO's Self Help Plus (SH+) and a session for Post-Migration Living Difficulties (PMLD) for Syrian women. SH+ is a guided self-help program with five weekly sessions led by facilitators, aimed at managing stress and psychological distress without requiring a diagnosis. This scalable intervention is based on solid research, proven effective in reducing stress and preventing mental health disorders (Tol et al., 2020; Turrini et al., 2019). The PMLD session, based on WHO's Problem Management Plus (PM+), involves focus groups to identify post-migration challenges. Participants share experiences, learn coping strategies, discover local resources, and strengthen social support networks. This integrated approach aims to enhance mental health, address post-migration difficulties, and improve stress reduction skills, supporting adaptation to a new country.
  Arms: Self Help Plus (SH+) combined with a session for Post Migration Living Difficulties (PMLD)

SUMMARY:
This study will conduct a two-arm, single-blind, randomized controlled trial among Syrian refugee women living in Turkey who experience psychological distress. In the study, participants will be randomly assigned to either the SH+ intervention (n = 105) combined with a session on Post-Migration Living Difficulties (PMLD) or Treatment as Usual (TAU) (n = 105). SH+ is a five-session guided self-help intervention focusing on stress management based on Acceptance and Commitment Therapy (ACT). In addition, a session discussing post-migration difficulties and possible problem-management techniques will be integrated after the SH+ intervention. This study aims to fill an important gap in refugee health and well-being research by focusing on the integrated expansion and implementation of an intervention program to address the psychosocial challenges faced by refugee Syrian women. The results will assess the effectiveness of the intervention on psychological distress, focusing on its potential positive effects on psychological distress, stress management, and adaptation processes. Furthermore, the impact of the intervention on the use of association services and psychological flexibility will be examined.

DETAILED DESCRIPTION:
The number of displaced people worldwide has reached 110 million, underscoring the urgent need to investigate and address the psychosocial effects of conflict and displacement. Syrian refugees, the largest displaced population, face significant mental health challenges, including heightened risks of Post-Traumatic Stress Disorder (PTSD), depression, and anxiety due to both traumatic experiences and post-migration stressors. The World Health Organization's (WHO) Self-Help Plus (SH+) intervention provides a valuable psychological support tool to help manage stress and mitigate these difficulties. Additionally, post-migration living difficulties, such as social integration issues, employment barriers, and cultural adaptation, critically affect asylum seekers' adjustment to new environments and their mental health. Addressing both the psychological and psychosocial aspects is crucial for effectively mitigating the complex challenges faced by asylum seekers, emphasizing the need for comprehensive support to improve integration and well-being in post-migration contexts.

This study will conduct a two-arm, single-blind, randomized controlled trial among Syrian refugee women living in Turkey who experience psychological distress. Participants will be randomly assigned to one of two groups: the SH+ intervention combined with a session on Post-Migration Living Difficulties (PMLD) or Treatment as Usual (TAU). Each group will consist of 105 participants, totaling 210 participants in the study. The SH+ intervention is a five-session guided self-help program based on Acceptance and Commitment Therapy (ACT), focusing on stress management. This intervention is designed to be accessible and does not require a diagnosis, making it suitable for a wide audience and particularly useful in areas with limited mental health services.

In addition to the SH+ intervention, the intervention group will participate in a session specifically addressing post-migration living difficulties. This session will occur after the completion of the SH+ intervention and will focus on identifying and managing challenges such as social integration, employment barriers, and cultural adaptation. Using problem-management techniques, this session aims to empower participants by enhancing their coping skills, building solidarity through shared experiences, and providing information about local resources available for asylum seekers. The integrated intervention aims to strengthen the mental health of the participants and provide comprehensive support for adapting to their new country.

The study will measure several outcomes to assess the effectiveness of the intervention. Primary outcomes include the reduction of psychological distress, measured using standardized tools such as Kessler Psychological Distress (K10). Secondary outcomes will focus on psychosocial traits. Additionally, the study will examine the impact of the intervention on the use of association services and psychological flexibility, which is a key component of ACT.

The intervention aims to fill an important gap in refugee health and well-being research by focusing on the integrated expansion and implementation of a comprehensive intervention program to address the psychosocial challenges faced by Syrian refugee women. By combining SH+ with a PMLD session, the study seeks to provide a holistic approach to improving the mental health and well-being of participants, offering them the necessary tools and knowledge to navigate the complexities of post-migration life. The results of this study are expected to provide valuable insights into the effectiveness of integrated psychosocial interventions and inform future efforts to support displaced populations globally.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (18 years and above),
* Selected among Syrian women residing in Turkey under temporary protection,
* Speak Arabic,
* Have not received any services from the Refugee Association before,
* A score of more than 16 on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0),
* A score of more than 15 on the Kessler-10 (K10) Psychological Distress Scale.

Exclusion Criteria:

* Have an acute medical condition,
* At risk of suicide,
* Have a severe mental disorder,
* Have severe cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is exclusively for women.
Enrollment: 210 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  Kessler Psychological Distress Scale (K10) The primary outcome measure of this study is the Kessler 10 (K10) scale developed by Kessler & Mroczek (2002). This scale is designed to measure general psychological distress experienced in the past 30 days without a specific cause. The scale was translated into Arabic and validated by Easton et al. (2017). This 10-item scale assesses each item using a 5-point Likert scale (1: Never; 5: Always). As a result of the reliability studies conducted for the Arabic translation of the scale, Cronbach's alpha (α) value was found to be .88 (Easton et al., 2017).

SECONDARY OUTCOMES:
Disability Assessment | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  WHO Disability Assessment Schedule (WHODAS 2.0) The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) is a 5-point Likert-type scale for general and clinical use, developed by Ustun et al. (2010) and validated by Akhtar et al. (2021) with a Cronbach's Alpha value of .74 for Arabic, and is designed to measure the disability of individuals.
Psychological Flexibility | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  The Acceptance and Action Questionnaire (AAQ-II) Within the scope of the study, the Acceptance and Action Questionnaire (AAQ-II) (Hayes et al., 2004) will be used to assess psychological flexibility. The translation of the scale into Arabic and validation study was conducted by Hemaid et al. (2016). The 7-item scale evaluates each item on a 7-point Likert scale (1: Never true; 7: Always true). As a result of the reliability studies conducted for the Arabic translation of the scale, Cronbach's Alpha (α) value was found to be .78 (Hemaid et al., 2016).
Symptoms of Post Traumatic Stress Disorder | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  PTSD Checklist for DSM-5 (PCL-5) The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) was developed by Weathers et al. (2013) as a 20-item 5-point Likert-type scale to measure PTSD symptoms and severity, and adapted into Arabic by Ibrahim et al. (2018) and gained validity and reliability with a Cronbach's Alpha value of .86.
Psychological Outcome Profiles | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  PSYCHLOPS PSYCHLOPS is a 6-point Likert-type scale with four and six items for pre and post-assessments, respectively, created by Ashworth et al. (2006) to assess individuals' psychological health conditions and the effects of their problems on their lives. The Arabic version has been used especially in studies on Syrian refugees (Acarturk et al., 2022; Uygun et al., 2020).
Well-being | Baseline, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  The World Health Organization- Five Well-Being Index (WHO-5) The WHO-5 Well-being Index is a short self-report rating scale developed by WHO (1998) to assess subjective well-being and general mental health condition and interest in the last two weeks on a 6-point Likert scale (0: Never; 5: Always). As a result of the Arabic validity and reliability study conducted by Alshayea (2023), it was found reliable with a Cronbach's alpha value of .91.
Post Migration Living Difficulties | Baseline, during the intervention, after the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  Post Migration Living Difficulties Checklist (PMLDC) The Post Migration Living Difficulties Checklist was developed by Silove et al. (1997) to measure post-asylum difficulties and related stress levels. It is a 17-item, 5-point Likert scale, the Arabic version of which has been used effectively in studies on forcibly displaced communities (Schick et al., 2016, 2018; Spaaij et al., 2023).
Service Uses | After the intervention (6 weeks after baseline), 3 months after the intervention, and 6 months after the intervention
  The study will include a service use inventory based on the Client Service Utilization Inventory (CSRI) (Beecham & Knapp, 1992) to assess the frequency and duration of use of association services by participants in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Keklik, Study Director — Medipol University
Locations (1):
- Refugees and Asylum Seekers Assistance and Solidarity Association (RASAS), Istanbul, Sultanbeyli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request and following the completion of the study, ensuring all necessary privacy and ethical guidelines are met. Interested researchers will need to submit a formal request and agree to use the data only for scientific purposes, adhering to any conditions set by the study's ethical committee and data-sharing policy.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD will be made available to other researchers starting from May 2025, following the completion of the study.
Access Criteria: Researchers requesting access to the IPD must submit a formal request detailing the purpose of their research and how they intend to use the data. Requests will be reviewed by the study's ethical committee to ensure compliance with privacy and ethical guidelines. Approved researchers will be required to sign a data use agreement, committing to use the data solely for scientific purposes, maintaining participant confidentiality, and adhering to all stipulated conditions.